CLINICAL TRIAL: NCT00597987
Title: BRCA1 Haploinsufficiency and Gene Expression
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Memorial Health University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 04-045
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: BRCA1 Mutations
Keywords: BRCA1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from cases will be collected from patients who have previously undergone genetic counseling through the Clinical Genetics Service at MSKCC and tested positive for a germline mutation in BRCA1. Blood samples from controls will be obtained from two sources.
  First from specimens already collected under IRB Protocol #99-030, entitled "Collection of Tissue, Blood, and Cells to be Used for Studying the Causes, Prevention, Diagnosis, and Treatment of Breast Cancer (T. King, PI). Controls will also be collected from patients who have previously undergone genetic counseling through the Clinical Genetics Service at MSKCC and tested negative for germline mutations in BRCA1. Isolation of total RNA from blood will be performed using the PAXgene™ Blood RNA System. This study will use lymphocyte RNA samples from 50 individuals with BRCA1 mutations and 50 age-matched controls. Gene expression profiling will be performed in the Genomics Core Laboratory of MSKCC.

GROUPS / COHORTS (1):
- 1: RNA samples

SUMMARY:
The purpose of this study is to collect a blood sample from patients that may be used for research purposes. These blood samples will be used by researchers at this institution to study the causes of breast and ovarian cancer, and to better understand how these cancers develop. We are trying to discover differences in the ways cells work in women with a high genetic risk of developing breast or ovarian cancer. Early data suggest that some genes may be turned on or off in different ways based upon whether or not a woman has a high genetic risk of developing breast or ovarian cancer. The primary objective is to test the hypothesis that BRCA1 haploinsufficiency regulates gene expression on the X chromosome. This hypothesis will be tested by comparing the gene expression profiles of BRCA1 heterozygotes (cases) to an age-matched group of unaffected women who are not BRCA1 mutation carriers (controls).

DETAILED DESCRIPTION:
The specific aim of this project is to test the hypothesis that BRCA1 haploinsufficiency regulates gene expression on the X chromosome. This hypothesis will be examined by determining if X chromosome gene expression profiles, derived from lymphocyte RNA, of BRCA1 mutation carriers (cases) can be distinguished from an age-matched group of women who do not have BRCA1 mutations (controls). Neither cases nor controls will have a history of cancer. This investigation will provide valuable insight into the biologic function of BRCA1 and its role in breast and/or ovarian tumorigenesis. Blood samples from cases will be collected from patients who have previously undergone genetic counseling through the Clinical Genetics Service at MSKCC and tested positive for a germline mutation in BRCA1. Blood samples from controls will be obtained from two sources.

First from specimens already collected under IRB Protocol #99-030, entitled "Collection of Tissue, Blood, and Cells to be Used for Studying the Causes, Prevention, Diagnosis, and Treatment of Breast Cancer (T. King, PI). Controls will also be collected from patients who have previously undergone genetic counseling through the Clinical Genetics Service at MSKCC and tested negative for germline mutations in BRCA1. Isolation of total RNA from blood will be performed using the PAXgene™ Blood RNA System. This study will use lymphocyte RNA samples from 50 individuals with BRCA1 mutations and 50 age-matched controls. Gene expression profiling will be performed in the Genomics Core Laboratory of MSKCC under the supervision of Agnes Viale, PhD. Class comparison analysis will be performed on the gene expression data in the Biostatistics Department under the supervision of Adam Olshen, PhD. It is anticipated that this study will be completed in approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

For acquisition of control specimens, samples already collected under IRB approved protocol 99-030 will be used. This protocol was a tissue and blood acquisition protocol entitled "Collection of Tissue, Blood, and Cells to Be Used for Studying the Causes, Prevention, Diagnosis, and Treatment of Breast Cancer". Patients have already given consent and signed a research authorization for to use their blood specimens for this purpose. Controls will also be collected from patients who have previously undergone genetic counseling through the Clinical Genetics Service at MSKCC and tested negative for a germline mutations in BRCA1. These individuals will be approached and asked to donate a sample at the time of their results appointment. Blood samples from cases will be collected from patients who have tested positive for a germline mutation in BRCA1. These women will have been participants in MSKCC protocols such as 96-51 and 97-29, or tested at outside institutions and receiving followup care at MSKCC. Any patient with a presumed pathogenic mutation in BRCA1 will be eligible for inclusion.

Exclusion Criteria:

Subjects will be eligible without regard to age, racial, or ethnic status. Subjects with any personal history of cancer will be excluded. Attending physicians authorized to obtain informed consent may exercise discretion in excluding individuals for appropriate medical or other (e.g., minors, mentally impaired) reasons. Patients with an unclassified variant in BRCA1 will be excluded as the functional significance of these variations is unknown.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be performed using lymphocyte RNA samples from 50 women with BRCA1 mutations and 50 age-matched controls without BRCA1 mutations. Class comparison analysis will be performed on the gene expression data.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2004-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The primary analysis of these data will be paired t-tests between the age-matched cases and controls for all genes on the X chromosome. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tari King, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org